CLINICAL TRIAL: NCT04724213
Title: Development and Validation of a Standardized Assessment Instrument for Health-related Quality of Life (HrQoL) in Children and Adolescents With Pompe Disease (PD): a Joint Effort of Patients, Caregivers and Metabolic Experts
Brief Title: Development of an Assessment Tool for Health-related Quality of Life in Children and Adolescents With Pompe Disease
Acronym: Pompe_HrQol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pompe_HrQol
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Testing of reliability / validity of new questionnaire (Other)
  Interventions: Other: Testing of reliability / validity of new questionnaire

INTERVENTIONS:
Other: Testing of reliability / validity of new questionnaire — Participants will answer new questionnaire and other, established, generic and chronic generic HrQol instruments

SUMMARY:
Health related quality of life (HrQoL), is "the patient's subjective perception of the impact of his disease and its treatment on his daily life, physical, psychological and social functioning and well-being" and thus constitutes a patient reported outcome (PRO) of utmost importance. Generic HrQoL instruments can by definition not capture disease-specific parameters nor are they sensitive enough to detect their changes. In this study, a disease-specific HrQoL questionnaire for children and adolescents will be developed. Patients and parents will be involved in focus groups and interviews to identify relevant contents. The instrument will be tested for validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD from age 8 years

  * Parent of patient(s) < 18 years with PD
  * Able to give informed consent as documented by signature
  * Sufficient command of the German language

Exclusion Criteria:

* - Inability to follow the procedures of the study, e.g. due to language problems or severely reduced health status

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Reliability/ validity of questionnaire | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Martina Huemer, Prof dr, Principal Investigator — University Childrens Hospital Zurich
Locations (1):
- University Childrens Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No